CLINICAL TRIAL: NCT06075147
Title: An Observational Study Program to Investigate the Effectiveness of Aflibercept 8 mg Used in DME and nAMD in a Real-world Setting
Brief Title: The SPECTRUM Study: An Observational Study to Learn More About How Well Aflibercept 8 mg Works in Treating Visual Impairment Due to Neovascular Age-related Macular Degeneration or Diabetic Macula Edema
Status: Active, not recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22480
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Visual Impairment; Neovascular Age-related Macular Degeneration (nAMD); Diabetic Macula Edema (DME)
MeSH Terms: conditions — Vision Disorders | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- naïve nAMD: Treatment-naive patients with nAMD
  Interventions: Drug: Aflibercept 8 mg (VEGF Trap-Eye, BAY86-5321)
- pretreated nAMD: Pretreated patients with nAMD
  Interventions: Drug: Aflibercept 8 mg (VEGF Trap-Eye, BAY86-5321)
- naïve DME: Treatment-naïve patients with DME
  Interventions: Drug: Aflibercept 8 mg (VEGF Trap-Eye, BAY86-5321)
- pretreated DME: Pretreated patients with DME
  Interventions: Drug: Aflibercept 8 mg (VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept 8 mg (VEGF Trap-Eye, BAY86-5321) — Following the manner of observational study, no intervention will be provided in the study. Any treatment decision, including the decision for aflibercept 8 mg treatment, is at the discretion of the attending physician, made in accordance with his/her experience and follows approved clinical guidelines.

SUMMARY:
This is an observational study in which only data are collected from people who have already been prescribed aflibercept 8 mg by their own doctors.

In this study, data from adults with visual impairment due to neovascular age-related macular degeneration (nAMD) or diabetic macula edema (DME) will be collected and studied.

Visual impairment is any degree of vision loss that affects a person's ability to perform daily activities. nAMD is an eye disorder that causes vision loss due to the growth of abnormal blood vessels that leak blood or retinal fluid into the macula (the central part of the retina). nAMD is a leading cause of vision loss for people aged 50 and older. DME is a diabetes-related eye disorder. In DME, the macula swells up due to fluid leakage from damaged blood vessels, resulting in vision problems.

Aflibercept 8 mg is a drug that is injected into the eye. It works by blocking a protein called vascular endothelial growth factor (VEGF) which causes abnormal growth and leakage of blood vessels at the back of the eye.

Aflibercept 8 mg has been submitted for approval for the treatment of visual impairment due to nAMD and DME based on the results from 2 studies called PHOTON and PULSAR. This study will begin once approval is obtained. Currently, no real-world data are available for aflibercept 8 mg.

The main purpose of this study is to collect more information about how well aflibercept 8 mg injection works in people with nAMD and DME. This study will include participants who have not received any prior treatment for nAMD or DME and participants who have.

The main information that researchers will collect:

the change in vision test scores called the best corrected visual acuity (BCVA) after 12 months of treatment.

Data will be collected from February 2024 to September 2027 and will cover a period of up to 24 months per participant. The data will be collected using medical records and by interviewing the patients during regular visits that take place in routine practice.

Researchers will observe participants from the first injection of aflibercept 8 mg until the end of the observation.

In this study, only available data from regular visits will be collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for patients with nAMD

* A diagnosis of nAMD
* Patient aged ≥50 years
* Patients for whom the decision to initiate treatment with intravitreal (IVT) aflibercept 8 mg according to a local product information was made as part of routine clinical practice
* Signed informed patient consent before the start of data collection (according to the requirements of the local authorities and laws)

Inclusion criteria for patients with DME

* A diagnosis of DME
* Patient aged ≥18 years (or country's legal age of adulthood if the legal age is >18 years) with type 1 or type 2 diabetes mellitus
* Patients for whom the decision to initiate treatment with IVT aflibercept 8 mg according to a local product information was made as part of routine clinical practice
* Signed informed patient consent before the start of data collection (according to the requirements of the local authorities and laws)

Exclusion Criteria:

Exclusion criteria for all patients with nAMD

* Participation in an investigational program with interventions outside of clinical routine practice
* Contraindications as listed in the local intravitreal aflibercept 8 mg local product information
* Extra/periocular infection or inflammation in either eye at time of first injection
* Patient receiving other intravitreal treatments other than aflibercept in the fellow eye
* Any medication interfering with aflibercept 8 mg in the intravitreal aflibercept 8 mg local product information Additional exclusion criteria for treatment-naïve patients with nAMD
* Any prior ocular treatment in the study eye or systemic treatment in nAMD Additional exclusion criteria for pretreated patients with nAMD
* Prior intravitreal anti-VEGF treatments in the study eye within the last 28 days
* Prior treatment with intravitreal corticosteroid in the study eye within the last 3 months
* Fluocinolone implant in the study eye within the last 3 years
* Dexamethasone implant in the study eye within the last 6 months
* Any concurrent drug releasing implant in the study eye

Exclusion criteria for all patients with DME

* Participation in an investigational program with interventions outside of clinical routine practice
* Contraindications as listed in the intravitreal aflibercept 8 mg local product information
* Extra/periocular infection or inflammation in either eye at time of first injection
* Patient receiving other intravitreal treatments other than aflibercept in the fellow eye
* Any medication interfering with aflibercept 8 mg in the intravitreal aflibercept 8 mg local product information
* Previous treatment of the study eye with laser in the last 90 days prior to first IVT aflibercept 8 mg Additional exclusion criteria for treatment-naïve patients with DME
* Any prior ocular treatment in the study eye or systemic treatment in DME Additional exclusion criteria for pretreated patients with DME
* Prior intravitreal anti-VEGF treatments in the study eye within the last 28 days
* Prior treatment with intravitreal corticosteroid in the study eye within the last 3 months
* Fluocinolone implant in the study eye within the last 3 years
* Dexamethasone implant in the study eye within the last 6 months
* Any concurrent drug releasing implant in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SPECTRUM will be performed in eye clinics and ophthalmology practices in several countries across North America, Europe, Middle East, and Asia Pacific.
  Female and male patients (aged ≥ 18 years for the DME cohorts or ≥ 50 years for the nAMD cohorts) with a diagnosis of nAMD or DME can be enrolled after the decision for treatment with aflibercept 8 mg has been made by the treating physician. Indications, contraindications, risks, warnings, and precautions according to the local market authorization/local product information should be carefully considered.
  For each patient a single eye will be considered as a study eye. The eye treated with aflibercept 8 mg will be considered as study eye. If treatment for both eyes is decided simultaneously, the study eye will be the worse eye as per discretion of the treating physician. Treatment of the 2nd eye will be considered as a concomitant treatment.
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
The change of best corrected visual acuity (BCVA) from baseline to 12 months as evaluated in routine clinical practice | At baseline and 12 months
  BCVA measurements at baseline (first injection of aflibercept 8 mg) and at 12 months as ETDRS letters (according to the Early Treatment Diabetic Retinopathy Study (ETDRS) chart or other methods (e.g. Snellen charts) used in the routine clinical practice in participating countries or sites (with conversion to ETDRS))

SECONDARY OUTCOMES:
The change of best corrected visual acuity (BCVA) from baseline to 4 weeks, 8 weeks, 6 months, and 24 months as evaluated in routine clinical practice | At baseline, 4 weeks, 8 weeks, 6 months and 24 months
Number of aflibercept 8 mg injections in the study eye during the first 6 months, the first year (12 months), the second year (24 months), and the entire observation period (last visit), respectively | Up to 24 months
  Performed intravitreal aflibercept 8 mg injections in study eye (including date)
Number of visits regarding the study eye by type of visit during the first 6 months, the first 12 months, and the 24 months treatment period | Up to 24 months
  Performed different type of visits for study eye
Number of treated study eyes with 5, 10, and 15 letters (or equivalent) BCVA gain/loss from baseline at 4 weeks, 8 weeks, 6, 12, and 24 months | At baseline, 4 weeks, 8 weeks, 6, 12 and 24 months
Change in central retinal thickness as measured by optical coherence tomography (OCT) from baseline to 4 weeks, 8 weeks, 6, 12, and 24 month follow up | At baseline, 4 weeks, 8 weeks, 6, 12 and 24 months
Number of participants with (serious) adverse events and (serious) drug-related adverse events | From the first application of aflibercept 8 mg up to 24 months

CONTACTS AND LOCATIONS:
Locations (18):
- Many Locations, Multiple Locations, Australia
- Many Locations, Multiple Locations, Canada
- Many Locations, Multiple Locations, Denmark
- Many Locations, Multiple Locations, Finland
- Many Locations, Multiple Locations, France
- Many Locations, Multiple Locations, Germany
- Many Locations, Multiple Locations, Italy
- Many Locations, Multiple Locations, Japan
- Many Locations, Multiple Locations, Netherlands
- Many Locations, Multiple Locations, Norway
- Many Locations, Multiple Locations, Portugal
- Many Locations, Multiple Locations, Saudi Arabia
- Many Locations, Multiple Locations, South Korea
- Many Locations, Multiple Locations, Spain
- Many Locations, Multiple Locations, Sweden
- Many Locations, Multiple Locations, Switzerland
- Many Locations, Multiple Locations, United Arab Emirates
- Many Locations, Multiple Locations, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.